CLINICAL TRIAL: NCT06558084
Title: Real-World Clinical Outcomes and Toxicity in Metastatic Breast Cancer Patients Treated With First or Second Line CDK 4/6 Inhibitors and Endocrine Therapy
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asmaa Ali, Assistant lecturer, Ain Shams University
Other Study IDs: CDKTOX2024
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Toxicity, Drug; Progression, Disease
Keywords: Breast cancer; CDK4/6 inhibitor; toxicity; PFS
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Disease Progression; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Metastatic breast cancer patients: metastatic breast cancer patient receiving CDK4/6i in 1st or 2nd line
  Interventions: Drug: CDK4/6 Inhibitor

INTERVENTIONS:
Drug: CDK4/6 Inhibitor — CDK4/6 inhibitor in first and second lines

SUMMARY:
To assess CDK4/6i toxicity and effect on PFS in the Egyptian population

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients aged 18 years old or more
* Female patients
* Histologically proven invasive breast cancer
* Histologically proven HR-positive and HER2-negative breast cancer
* Metastatic breast cancer (Stage 4 according to AJCC 8th edition 2017)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 3.
* Adequate hematological and organs function
* Patients receiving CDK 4/6 inhibitor combined with endocrine therapy(Aromatase inhibitors , GnRH agonists, fulvastrent). as a first or second line treatment

Exclusion Criteria:

* - Male breast cancer patients
* Patients in, visceral crisis (defined as : severe organ dysfunction, as assessed by signs and symptoms, laboratory studies and rapid progression of disease ) that are at risk of life threatening complication in the short term.
* Prior treatment with any CDK 4/6 inhibitor.
* History of any other cancer , unless in complete remission with no therapy for a minimum of 3 years.
* Have active bacterial or fungal infection, or detectable viral infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Breast Cancer patients attending Ain Shams University Clinical Oncology and Nuclear Medicine Department breast clinic from July 2022 till December 2024
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Adverse effect | 2 years
  assess the toxicity profile

SECONDARY OUTCOMES:
PFS | 2 years
  PFS in patient receiving CDK4/6i in Egypt

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University, Cairo, Egypt